CLINICAL TRIAL: NCT04481646
Title: The Efficacy and Feasibility of Face Mask Sampling for Hospitalised Adult Patients and Healthcare Workers With Suspected COVID-19
Brief Title: Novel Face Mask Sampling for COVID-19: A Diagnostic and Public Health Tool
Acronym: COVMASK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0775
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Biospecimen Retention: Samples With DNA — Face mask sample (exhaled sample)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients admitted to hospital with COVID-19 symptoms will be approached to undertake a face mask sample and nasopharyngeal swab at two time points 12 hours apart on a single day whilst in hospital. Medical records will be accessed for basic clinical, demographic and microbiological data.
  Interventions: Diagnostic Test: Face mask sampling
- 2: Healthcare workers who have report COVID-19 symptoms will be asked to undertake a face mask sample and nasophayngeal swab on days 1,3,5,7,10,14 and 21 of the study, for part of which they will be quarantined at home.During this time they will complete a simple symptom diary. Medical records will be accessed for basic clinical, demographic and microbiological data.
  Interventions: Diagnostic Test: Face mask sampling
- 3: Healthcare workers from different areas of the hospital will be approached as part of a screening programme. They will be asked to undertake a single face mask and swab sample. Basic clinical and environmental data will be collected about each participant so they exposure risk can be stratified.
  Interventions: Diagnostic Test: Face mask sampling

INTERVENTIONS:
Diagnostic Test: Face mask sampling — Mask sampling consists of a modified face mask (flat surgical, duckbilled or FFP1) which contains up to strips of 3D printed Polyvinyl alcohol (PVA). As outlined in our previous work (ref lancet). These PVA strips are manufactured by the University of Leicester and measure approximately 50mm x 500mm and are fixed into place by adhesive pads. Mask assembly is conducted at the University of Leicester and are sterilised prior to use. Figure 3 and 4 shows examples of the inside of the mask with 4 strips placed inside and of how it is worn by study participants. The mask sampling system has been approved for previous studies in the UK, South Africa and The Gambia and has current approval for service improvement work at University Hospitals of Leicester NHS Trust for respiratory pathogens. It is awaiting approval as a medical device with the Medicines and Healthcare products Regulatory Agency.

SUMMARY:
COVID-19 has become a global problem. There is an urgent need to improve the diagnosis and screening of patients and healthcare workers for COVID-19 in the UK. Mask based sampling is a method of detecting SARS-COV-2 (the virus responsible for COVID-19) in the breath of suspected COVID-19 patients or healthcare workers in the mask that they would wear in hospital. The investigators have previously demonstrated the utility of this method in other respiratory infections, such as tuberculosis.

This project aims to investigate the utility of mask-based sampling is a tool for the diagnosis and quantification of COVID-19 in breath and the implications in a healthcare setting using three cohorts of participants. Initially we will compare the amount of COVID-19 detected by mask sampling compared with standard nasopharyngeal swab, which is the current gold standard test, in patients who present to hospital with COVID-19 symptoms.

We will address the length of time COVID-19 is breathed out by people affected by the virus and the how infectious the virus is over time in a cohort of symptomatic healthcare workers who are isolating at home. This will allow us to understand how long someone stays infectious for and may have the potential to inform public health measures, for instance when healthcare workers can return to work or duration of isolation. Finally we will investigate asymptomatic carriage of COVID-19 by different healthcare workers in different areas of the hospital during a screening study. This will allow us to understand the extent of infection amongst healthcare workers and allow us to address hospital acquired transmission.

DETAILED DESCRIPTION:
In order to understand the utility of face mask sampling for the diagnosis of COVID-19 and the public health implications, three cohorts of participants will be asked to take part in this study. Each participant will be asked to wear a modified face mask containing strips of sampling material for up to one hour and undertake a nasopharyngeal (nose/throat) swab concurrently. Depending on which cohort the participants are recruited to, the number of these 'sampling sessions' will vary. Basic demographic and microbiological data will be collected for every participant.

Cohort 1:

Patients admitted to hospital with COVID-19 symptoms will be approached to undertake a face mask sample and nasopharyngeal swab at two time points 12 hours apart on a single day whilst in hospital. Medical records will be accessed for basic clinical, demographic and microbiological data.

Cohort 2:

Healthcare workers who have report COVID-19 symptoms will be asked to undertake a face mask sample and nasophayngeal swab on days 1,3,5,7,10,14 and 21 of the study, for part of which they will be quarantined at home.

During this time they will complete a simple symptom diary. Members of the research team will visit their home to consent and train them on sampling techniques on day 1. Masks and swabs will then be left with them to complete.

These samples will then be collected at a mutually convenient time as teh samples are sample at room temperature for many days. If the healthcare worker does not feel able to complete self-sampling then a research team member will visit to undertake the sampling. Full PPE will be worn at all times and Staff working on the study will have NHS honorary contracts in place and will operate under University Hospitals of Leicester NHS Trust policies and procedures surrounding infection control and risk assessments whilst conducting this research. Medical records will be accessed for basic clinical, demographic and microbiological data. The results of the face mask sample are not intended to provide any diagnostic results and as such, the results will not be made available to the participant or the Occupational Health Department and HCWs will be directed to continue to follow the University Hospitals of Leicester NHS Trust policy when determining whether or not they are safe and able to return to work.

Cohort 3:

Healthcare workers from different areas of the hospital will be approached as part of a screening programme. They will be asked to undertake a single face mask and swab sample. Basic clinical and environmental data will be collected about each participant so they exposure risk can be stratified. The research team will work closely with the senior managers of each area to introduce the study to each participant so to minimise any stigmata related to deciding to participate or not. Any participant that has either a mask or swab positive result will be followed up and offered conventional screening as per Public Heath England's guidance. Staff working on the study will have NHS honorary contracts in place and will operate under University Hospitals of Leicester NHS Trust policies and procedures surrounding infection control and risk assessments whilst conducting this research. HCWs will be reminded that the results of the FSM are not conclusive and should not be used for diagnostic purposes. Each individual who produces a FSM+ sample will be referred back to the Trust Occupational Health Department for followup and management as per Trust policy.

ELIGIBILITY:
Inclusion Criteria:

* Not requiring oxygen by face mask
* Either:

  o Patients admitted to hospital with suspected COVID-19
* Or o Healthcare workers working within University Hospitals of Leicester, including those with and without symptoms suspicious of COVID-19.

Exclusion Criteria:

* Participants requiring oxygen by face mask (i.e., Venturi, non rebreathe)
* Participants with respiratory failure
* Medical history that might, in the opinion of the attending clinician, put the patient at significant risk if he/she were to participate in the study
* Individuals who are unable to provide informed consent for themselves (i.e., individuals who lack capacity).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: as previously described
Sampling Method: Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparison with Naso-pharyngeal swab | 6 months
  Newly diagnosed patients compare mask and swab samples taken at the same time
Mask out over time | 12 months
  SARS-COV-2 RNA quantification over time SARS-COV-2 RNA quantification over 21 days post diagnosis
mask as a screening tool in asymptomatic people | 6 months
  screening of asymptomatic healthcare workers

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided